CLINICAL TRIAL: NCT02382341
Title: A Radiographic Study of Patients Treated With the BIOSURE™ HEALICOIL™ PK Interference Screw for ACL Repair With Soft Tissue Fixation
Brief Title: BIOSURE™ HEALICOIL™ PK Bone In-growth Study
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 15000946
Record Dates: First submitted 2015-02-13; First posted 2015-03-06 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2017-04

CONDITIONS: Deficiency of Anterior Cruciate Ligament
Keywords: ACL; BIOSURE; HEALICOIL; PEEK; In-Growth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: BIOSURE™ HEALICOIL™ PK Interference Screw
  Interventions: Device: BIOSURE™ HEALICOIL™ PK Interference Screw

INTERVENTIONS:
Device: BIOSURE™ HEALICOIL™ PK Interference Screw — Subjects will receive the appropriate sized BIOSURE™ HEALICOIL™ PK Interference Screw

SUMMARY:
The study seeks to document the bone in-growth into the BIOSURE™ HEALICOIL PK screw as measured by CT scans. Patients' improvement in pain and function will also be followed through various outcome measures.

DETAILED DESCRIPTION:
The primary objective of the current study is to assess bone in-growth in the BIOSURE™ HEALICOIL™ Interference screw in the tibial tunnel of patients undergoing ACL reconstruction with soft tissue grafts; tunnel widening and change in IKDC knee and subjective scores will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* ACL tear requiring surgical reconstruction with semitendinosus/gracilis graft.
* Willing and able to give voluntary informed consent to participate in this study
* Willing and able, in the opinion of the investigator, to cooperate with study procedures and willing to return to study site for all post-operative study visits.
* Subject is between 18 and 50 years at the time of surgery
* ASA group 0-2 (limited medical illness).

Exclusion Criteria:

* Revision ACL reconstruction
* Cartilage injury (IKDC Grade IV lesion> 2 cm2)
* Current malignant disease
* Rheumatoid arthritis
* Osteonecrosis or Avascular Necrosis
* Ankylosing spondylitis
* Subject is Obese; BMI > 35
* Subject is pregnant or plans to become pregnant during the study
* Subject has received medical treatment within 6 weeks of enrollment with any of the following:

Glucocorticoids Growth hormone

* Participating in another investigational trial or on-going study that would interfere with the assessment of the primary and secondary outcomes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing ACL reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-09-12 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Bone In-growth measured by CT scans | 1 year
  Bone In-growth measured by CT scans

SECONDARY OUTCOMES:
Bone In-growth measured by CT scans | 6 months
  Bone In-growth measured by CT scans
Improvement in IKDC Knee Examination scoring from baseline to 1 year post-operatively | 1 year
Improvement in the IKDC Subjective Knee Evaluation scoring from baseline to 1 year post-operatively | 1 year
Improvement in IKDC Knee Examination scoring from baseline to 2 years post-operatively | 2 years
Improvement in the IKDC Subjective Knee Evaluation scoring from baseline to 2 years post-operatively | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lind, MD, PhD, Principal Investigator — Aarhus University Hospital

REFERENCES:
- [Derived] Lind M, Nielsen T, Sorensen OG, Mygind-Klavsen B, Fauno P, Leake-Gardner S. Bone ingrowth into open architecture PEEK interference screw after ACL reconstruction. J Exp Orthop. 2020 Sep 18;7(1):68. doi: 10.1186/s40634-020-00285-z. PMID 32948982